CLINICAL TRIAL: NCT04899986
Title: Clinical Comparison Between Chlorhexidine Gel and Peribioma Periogel in Patients With Peri-implant Mucositis: a Split-mouth Randomized Clinical Trial.
Brief Title: Chlorhexidine Gel and Peribioma Periogel Use in Peri-implant Mucositis Sites: a Split-mouth Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-PBIMPLANT
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Peri-implant Mucositis
Keywords: non-surgical periodontal therapy
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): Patients from this group will use chlorhexidine Biorepair gel and toothpaste for home oral care.
  Interventions: Other: Chlorhexidine and Biorepair gel and toothpaste application
- Control Group (Active Comparator): Patients from this group will not use chlorhexidine and Biorepair gels and toothpastes, but will perform home oral care with standard toothpastes.
  Interventions: Other: Standard oral hygiene

INTERVENTIONS:
Other: Chlorhexidine and Biorepair gel and toothpaste application — Split-mouth application of chlorhexidine gel 1% (quadrants 1 and 4) and Biorepair Periogel (quadrants 2 and 3) after professional dental hygiene. Home oral care will be continued with chlorhexidine 0,12% gel and Biorepair Periogel in the same quadrants, for the following 15 days from the visits, together with the use of Biorepair Parodontogel toothpaste.
  Arms: Trial Group
Other: Standard oral hygiene — Use of standard toothpastes for home oral hygiene.
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the efficacy of non-surgical periodontal therapy with supportive home oral care for the treatment of peri-implant mucositis.

Patients with bilateral implants with peri-implant mucositis will undergo professional dental hygiene with ultrasonic handpiece and manual scaler, followed by the application of glycine Airflow powders. Then, patients will be randomly divided into two groups: the Trial Group will undergo a split-mouth application of chlorhexidine gel 1% for quadrants 1 and 4 and of Biorepair Periogel 0.12% for quadrants 2 and 3, with one daily home application for the following 15 days after the visits and the use of Biorepair Parodontogel toothpaste; the control Group will not use any gels.

The improvement of peri-implant mucositis will be evaluated between the two groups and differences between the two gels will be assessed, if present.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of non-surgical periodontal therapy with supportive home oral care for the treatment of peri-implant mucositis.

Patients with bilateral implants with peri-implant mucositis will undergo professional dental hygiene with ultrasonic handpiece and manual scaler, followed by the application of glycine Airflow powders. Then, patients will be randomly divided into two groups:

* Trial Group: split-mouth application of chlorhexidine gel 1% for quadrants 1 and 4 and of Biorepair Periogel 0.12% for quadrants 2 and 3. Home oral care will be continued with 1 application per day of the two gels for the following 15 days after the visits for the same quadrants, and the use of Biorepair Parodontogel Toothpaste.
* Control Group: no application neither of chlorhexidine gel nor of Biorepair Periogel.

The improvement of peri-implant mucositis will be evaluated between the two groups and differences between the two gels will be assessed, if present, evaluating periodontal indices at the baseline, after three months and after six months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-70 years)
* Bilateral presence of peri-implant mucositis
* Patients with high compliance

Exclusion Criteria:

* Patient with cardiac pacemaker
* Patients suffering from psychological, neurological or psychiatric disorders
* Patients suffering from systemic, metabolic or autoimmune diseases
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Change in BOP - Bleeding On Probing | Baseline, 1, 3 and 6 months.
  Dichotomous scoring (yes/no)
Change in GBI - Gingival Bleeding Index (percentage) | Baseline, 1, 3 and 6 months.
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  The number of bleeding sites is divided per the total number of probed sites; the ratio is multiplied X 100.
Change in suppuration | Baseline, 1, 3 and 6 months.
  Dichotomous scoring (yes/no)
Change in marginal mucosa condition | Baseline, 1, 3 and 6 months.
  Scoring criteria:
  * 0: normal mucosa
  * 1: minimal inflammation with color change and minor edema
  * 2: moderate inflammation with redness, edema and glazing
  * 3: severe inflammation with redness, edema, ulceration and spontaneous bleeding without probing
Change in mucosal margin | Baseline, 1, 3 and 6 months.
  Dichotomous scoring (migrated/non migrated)
Probing Pocket Depth | Baseline, 1, 3 and 6 months.
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in PI - Plaque Index (percentage) | Baseline, 1, 3 and 6 months.
  Evaluation of the presence of plaque on the 4 surfaces of teeth on the total amount of dental surfaces.
Change in BS - Bleeding Score | Baseline, 1, 3 and 6 months.
  Scoring criteria:
  * 0: no bleeding
  * 1: isolated visible spots
  * 2: blood forms a confluent red line on mucosal margin
  * 3: heavy or profuse bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator